CLINICAL TRIAL: NCT04365751
Title: A Prospective Multicenter Cohort Control Study of Percutaneous Microwave Ablation and Laparoscopic Resection for Hepatocellular Carcinoma With a Diameter of 3.1 ~ 5.0cm
Brief Title: To Compare the Efficacy of Microwave Ablation and Laparoscopic Hepatectomy for Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Interventional ultrasound department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019002
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: microwave ablation, hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous microwave ablation group (Experimental): MWA (Microwave) is an ultrasound-guided, minimally invasive technique that implants ablation electrodes into target tissue to rapidly generate high temperatures and rapidly develop coagulative necrosis in tumor tissue, thereby achieving the goal of local tumor treatment.
  Interventions: Procedure: Percutaneous microwave ablation, Laparoscopic hepatectomy
- Laparoscopic hepatectomy (Other): Laparoscopic hepatectomy is a widely used surgical technique in the treatment of benign (malignant) liver diseases
  Interventions: Procedure: Percutaneous microwave ablation, Laparoscopic hepatectomy

INTERVENTIONS:
Procedure: Percutaneous microwave ablation, Laparoscopic hepatectomy — For patients with hepatocellular carcinoma who meet the enrollment requirements, under the guidance of ultrasound, microwave ablation electrodes were implanted into the tumor tissues by percutaneous puncture, and the high-temperature heat energy was generated to cause coagulation necrosis of the tumor, so as to achieve the goal of local tumor treatment with minimally invasive technology.

SUMMARY:
The study was a prospective multicenter cohort control study, which was divided into 1:1 groups to compare the clinical efficacy of percutaneous microwave ablation and laparoscopic hepatocellular carcinoma resection (tumor diameter 3.1-5.0cm).

DETAILED DESCRIPTION:
Research objectives:

To compare the clinical efficacy of percutaneous microwave ablation and laparoscopic resection for hepatocellular carcinoma (tumor diameter 3.1-5.0cm).

Research background:

Liver cancer is the sixth most common tumor in the world and the second leading cause of death. Due to the hepatitis B epidemic, the incidence of liver cancer in China is very high, accounting for about half of the global statistics on the number of new liver cancer cases and deaths each year. Current treatment guidelines recommend surgical resection or transplantation as the gold standard for the treatment of very early or early HCC patients. Meanwhile, local ablation is gradually accepted by clinicians for its minimally invasive nature, safety and efficacy, and it is recommended as an alternative treatment for tumors within 3cm. However, the choice of treatment for 3.1-5cm HCC based on a number of current retrospective studies is controversial. Therefore, we designed this study to provide reliable prospective data to support the selection of therapeutic modalities for HCC.

Technical introduction:

Microwave ablation (MWA) is an ultrasound guided ablation electrode implanted in the target tissue, in the form of electromagnetic waves to generate microwave energy, microwave can make the surrounding tissue in the water molecules oscillate against the friction of heat, high temperature heat causes rapid coagulation necrosis of the tissue, so as to achieve the purpose of local tumor treatment. Compared with other ablation techniques, MWA in the treatment of solid tumors can achieve higher tumor internal temperature in a shorter period of time, with strong penetration, synergistic effect of multi-needle combined ablation, and little influence by carbonization and blood perfusion. Therefore, MWA has fast heat production, high intracellular temperature, short ablation time and large ablation range.

Laparoscopic liver resection (Laparoscopic hepatectomy) reported for the first time in 1991 by the professor Reich. Laparoscopic techniques in the application in benign (malignant) liver disease is widespread. In China, since professor Weiping Zhou and others completed the first laparoscopic liver resection in mainland China in 1994, there have been continuous literature reports, and the scope and difficulty of surgical resection have been increasing.The 2008 Louisville declaration states that laparoscopic liver surgery is safe and effective for surgeons with extensive experience in hepatobiliary surgery and laparoscopic surgery.

Research methods In this study, 1134 patients were expected to be enrolled according to the 1:1 grouping of the experimental group and the control group. The efficacy of the two treatment methods was evaluated by comparing the overall survival of the two groups and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* 1.Older than 18 years old, regardless of gender; 2.In patients without cirrhosis background, hepatocellular carcinoma was definitely pathologically diagnosed within 1 month before surgery. In patients with cirrhosis background, dynamic contrast enhanced MRI/ multi-stage dynamic enhanced CT were used to determine the characteristic vascular signs of primary liver cancer (rapid heterogeneous vascular enhancement in arterial phase, rapid elution in venous phase or delayed phase); 3.The number of tumors was ≤3, and the maximum diameter of at least one tumor was 3.1-5.0cm; 4.No vascular and lymph node invasion and distant metastasis; 5.Liver function: child-pugh A or B (assessed within 14 days before surgery); 6.Subjects will understand the purpose of the study, voluntarily participate and sign the informed consent.

Exclusion Criteria:

* 1.Severe hepatic decompensation, presence of hepatic encephalopathy, massive ascites or gastrointestinal bleeding within 1 month; 2.Clotting disorders or bleeding tendencies (platelet count <50 x 109 / L or INR>1.5); 3.Patients with severe cardiac, pulmonary and renal insufficiency; 4.Combined with active infection; 5.Pregnant patients; 6.A history of drug abuse and mental illness; 7.Inability to tolerate pneumoperitoneum; 8.Other studies or anti-tumor therapists in the first four weeks of the study; 9.The researchers determined that there were any other factors that were inappropriate for inclusion or that affected participants' participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 60 months
  Defined as the length of time from the beginning of treatment to death or the last follow-up (if no death).

SECONDARY OUTCOMES:
Progression-free survival | 60 months
  Defined as the period of time between the time the patient is treated and the time the disease progresses or death from any cause is observed
Intrahepatic recurrence rate | 60 months
  Defined as the proportion of patients with intrahepatic recurrence from the beginning of the study to the end of the study or the death of the patients
Rate of extrahepatic metastasis | 60 months
  Defined as the proportion of cases with extrahepatic metastasis from the beginning of the study to the end of the study or the death of the patient
Local rate of progression | 60 months
  Defined as the proportion of patients with active tumor at the edge of the treatment area during follow-up after the tumor was completely treated

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No